CLINICAL TRIAL: NCT04316715
Title: Evaluation of Life-Steps to Enhance Adherence and Engagement in PrEP Care
Brief Title: Life-Steps Counseling to Enhance Adherence and Engagement in PrEP Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven Safren, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20190646; R01MH118043 (NIH)
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Adherence, Medication
Keywords: Life-Steps; HIV Prevention
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Life-Steps for PreP (Experimental): Participants in this group will receive standard of care treatment plus daily text message reminders. A subset of participants who demonstrate continued adherence challenges will also receive 4-6 weekly sessions of the Lifesteps for PrEP intervention.
  Interventions: Behavioral: Lifesteps for PrEP; Behavioral: Daily text message reminders
- Standard of Care (No Intervention): Participants in this group will not receive an intervention outside the standard of care.

INTERVENTIONS:
Behavioral: Lifesteps for PrEP — Four weekly nurse delivered counseling sessions plus two optional booster sessions. Sessions last approximately 40-50 minutes each. Sessions employ cognitive behavioral (CBT) techniques, motivational interviewing (MI), and psychoeducation.
  Arms: Life-Steps for PreP
Behavioral: Daily text message reminders — Participants get daily text messages on their cell phone reminding them to take their PrEP medication.
  Arms: Life-Steps for PreP

SUMMARY:
The purpose of this study is to test how different types of interventions may affect how someone takes their pre-exposure prophylaxis (PrEP) medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older
2. Male sex at birth or trans man (current gender identity is male) assigned female sex at birth
3. Self-reports as a person who has sex with men
4. PrEP naïve or is currently prescribed PrEP and reports uncertainty about future adherence
5. Medical providers at each site will determine that the participant is indicated for PrEP per Centers for Disease Control (CDC) guidelines
6. Screens in for currently having one or more of the following psychosocial syndemic problems: depression; heavy alcohol use; problematic substance use or polydrug use; history of trauma or abuse; and/or current interpersonal violence
7. Owns a cell phone that has texting and internet / data capacity

Exclusion Criteria:

1. Unable to provide informed consent due to severe mental or physical illness, cognitive impairment, or substance intoxication at the time of interview
2. Discovery of active suicidal ideation or major mental illness (e.g. untreated psychosis or mania) at the time of enrollment (these patients will be referred immediately for treatment, but may join the study when this is resolved)
3. Laboratory or clinical findings that would preclude PrEP initiation (e.g. decreased creatinine clearance)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
TFV-DP concentrations | 3, 6, 9, 12, 15, and 18 months
  Medication adherence as reported by Tenofovir diphosphate (TFV-DP) concentrations measured using dried blood spot (DBS) testing.
Wilson Medication Adherence self-report | up to 18 months
  Medication adherence as reported by the Wilson Medication Adherence self-report. The questionnaire has a total score ranging from 0-40, with a higher score indicating greater adherence.

SECONDARY OUTCOMES:
Retention in PrEP care | 3, 6, 9, 12, 15, and 18 months
  The percentage of participant attendance at follow up visits over 18 month study participation

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Safren, Ph.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Fenway Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No